CLINICAL TRIAL: NCT00002013
Title: A Safety, Pilot Pharmacokinetics and Neurocognitive Study of AS-101 in Combination With Zidovudine in AIDS/ARC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 045C; 753A-109-US
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; ammonium trichloro(dioxoethylene-O,O'-)tellurute; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; ammonium trichloro(dioxoethylene-O,O'-)tellurate

INTERVENTIONS:
Drug: Zidovudine
Drug: AS-101

SUMMARY:
To evaluate safety, pharmacokinetics, immunologic parameters and neurocognitive data for three dosages of AS-101 in combination with zidovudine (AZT) in patients with AIDS or AIDS related complex (ARC).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Zidovudine (AZT).
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Allowed ONLY with permission of the Wyeth-Ayerst medical monitor:
* Standard therapy for infections that develop during the study period.
* Oral acyclovir.
* Nystatin.
* Ketoconazole.
* Immunomodulators.
* Specific therapy for malignancies (including Kaposi's sarcoma).

Patients must have the following:

* Diagnosis of AIDS or AIDS related complex (ARC).
* Provide informed written consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection or malignancy requiring treatment at study entry.
* Prior history of psychiatric illness or head injury which in the judgment of the neuropsychologist would impair interpretation of the neurocognitive data.
* Evidence of central nervous system (CNS) opportunistic infection or malignancy.
* Serious underlying medical problems, including insulin- dependent diabetes mellitus, unstable ASHD (atherosclerotic heart disease) or uncontrolled hypertension, which may complicate interpretation of treatment results.
* Dementia.
* Evidence of = or > 2 + proteinuria at study entry.

Concurrent Medication:

Excluded without permission of the Wyeth-Ayerst medical monitor:

* Immunomodulators.
* Specific therapy for malignancies (including Kaposi's sarcoma).

Patients with the following are excluded:

* Active opportunistic infection or malignancy requiring treatment at study entry.
* Prior history of psychiatric illness or head injury which in the judgment of the neuropsychologist would impair interpretation of the neurocognitive data.
* Evidence of conditions listed in the Patient Exclusion Co-existing Conditions.
* Active substance abuse.
* Unlikely or unable to comply with the requirements of the protocol.

Prior Medication:

Excluded within 8 weeks of study entry:

* Immunomodulators.
* Antiviral therapy, except zidovudine.
* Excluded within 2 weeks of study entry:
* Intravenous or oral acyclovir.
* Excluded within 3 months of study entry:
* Ribavirin.

Required:

* Zidovudine at a dose of = or > 1000 mg/day for at least 6 weeks prior to study entry.

Active substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County - USC Med Ctr, Los Angeles, California, United States

REFERENCES:
- [Background] Laporate JP, Frottier J, Dormont D, Imbert JC, Albeck M, Najman A. As 101 in association with azt in AIDS patients: a phase I pilot study. Int Conf AIDS. 1989 Jun 4-9;5:405 (abstract no WBP320)